CLINICAL TRIAL: NCT02949596
Title: Prospective Cohort on Quality of Sexual Life Among Men Who Have Sex With Men Treated for Anal Cancer With Concurrent Chemotherapy and Intensity-modulated Radiotherapy
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Geovanne Pedro Mauro, MD, Instituto do Cancer do Estado de São Paulo
Other Study IDs: 576/15
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Anal Cancer; Quality of Life
Keywords: quality of sexual life; intensity-modulated radiotherapy; concurrent chemoradiotherapy
MeSH Terms: conditions — Anus Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Quality of life and quality of sexual life questionnaires

SUMMARY:
Treatment of anal cancer has been always linked to quality of life. Recently, with development on radiotherapy technique, toxicities have been lowered with the maintenance of adequate rates of disease control. This trial intends to follow patients prospectively with questionnaires to evaluate sexual quality of life among patients who are who men who have sex with other men and have been subject to concurrent chemoradiotherapy with IMRT technique.

DETAILED DESCRIPTION:
In this prospective single-arm cohort, patients who are men who have sex with other men will be recruited to answer routine questionnaires on quality of life in general and sexual quality of life in specific, most validated and other waiting for validation in Portuguese language. These questionnaires will be applied after the diagnose and before the beginning of the treatment, on the last day of treatment, and 3, 6 and 12 months after the treatment is completed. Only patients who will be treated with concurrent chemotherapy will be recruited, and intensity-modulated radiotherapy technique is mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Anal cancer proven biopsy
* men who have sex with other men
* curative intent of treatment
* IMRT required
* concurrent chemotherapy required

Exclusion Criteria:

* Patients who have undergone surgery for anal cancer
* patients who can't read, write or are unable to answer to questionnaire

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with anal cancer who are men who have sex with other men and are able to answer to questionnaires
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-10; Primary Completion 2020-10 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Evaluate quality of life validated questionnaire (EORTC QLQ-30) among patients treated for anal cancer with concurrent chemoradiotherapy who are men who have sex with other men | 2015-2020
Evaluate quality of life validated questionnaire (SF-36) among patients treated for anal cancer with concurrent chemoradiotherapy who are men who have sex with other men | 2015-2020
Evaluate quality of sexual life validated questionnaire (IIEF) among patients treated for anal cancer with concurrent chemoradiotherapy who are men who have sex with other men | 2015-2020

SECONDARY OUTCOMES:
Evaluate quality of sexual life with other questionnaires (CSFQ-14) that are not validated in Portuguese language in the same population | 2015-2020
Evaluate quality of sexual life with other questionnaires (ISL) in the same population | 2015-2020
Evaluate quality of sexual life with other questionnaires (MSHQ-short version) in the same population | 2015-2020
Evaluate quality of sexual life with other questionnaires (SEAR) in the same population | 2015-2020
Evaluate quality of sexual life with other questionnaires (SEX-Q) in the same population | 2015-2020
Evaluate quality of sexual life with other questionnaires (SHIM) in the same population | 2015-2020
Evaluate quality of sexual life with other questionnaires (CAYA-t) in the same population | 2015-2020
Evaluate quality of life among patients who are HIV positive in this cohort with the use of questionnaire HAT-QoL | 2015-2020

CONTACTS AND LOCATIONS:
Overall Officials: Geovanne Mauro, MD, Principal Investigator — physician
Locations (1):
- ICESP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No